CLINICAL TRIAL: NCT00307268
Title: Evaluating Clinical Outcomes of Treatment Effectiveness for Children and Adolescents With ADHD: An Observational, Long-Term Follow-up Study of Routine Clinical Care
Brief Title: Evaluating Clinical Outcomes of Treatment Effectiveness for Children and Adults With ADHD
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Eli Lilly and Company (Industry); Janssen-Ortho LLC (Industry); Purdue University (Other); Shire (Industry)
Responsible Party: Sponsor
Other Study IDs: H05-70361
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD Effectiveness
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate clinical effectiveness of medication treatment for ADHD. It is hypothesized that the effectiveness is lower than efficacy outcomes measured in clinical trials

DETAILED DESCRIPTION:
This is a prospective, long-term, observational study of routine clinical care. The study measurements will be integrated into the clinical assessment and follow-up procedures of the outpatient services under the Provincial ADHD Program. The study is designed for systematic follow-up of children and adolescents, diagnosed with ADHD irrespective of comorbidity or whether they elect to receive medication treatment. Evaluations occur every 6 months for 24 months. The population to be examined is children and adolescents with a diagnosis of ADHD, aged 6 to 18 inclusive (at baseline), referred to the Provincial ADHD Program for clinical assessment. No studies have been conducted that have evaluated the outcome of core ADHD symptoms in a clinic setting. Metaanalysis of clinical trials of medication treatment for ADHD have suggested an effect size of approximately 0.8. Because of the heterogeneity of the clinic sample, a much lower effect size can be anticipated. Two hundred patients will be enrolled in this study with primary measure of effectiveness being change in ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

Meet DSM-IV criteria for ADHD

Exclusion Criteria:

None

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents with a diagnosis of ADHD, aged 6 to 18 inclusive (at baseline), referred to the Provincial ADHD Program for clinical assessment.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Weiss, MD, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- Children's and Women's Health Centre of BC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Craig SG, Weiss MD, Hudec KL, Gibbins C. The Functional Impact of Sleep Disorders in Children With ADHD. J Atten Disord. 2020 Feb;24(4):499-508. doi: 10.1177/1087054716685840. Epub 2017 Jan 16. PMID 28093033